CLINICAL TRIAL: NCT04469777
Title: Evaluation of the Effect of Subcutaneous Injection of Erythropoietin on Visual Functions in Patients With Late Onset Optic Neuropathy
Brief Title: Subcutaneous Injection of Erythropoietin on Visual Functions in Patients With Late Onset Optic Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Fahmy Doheim, Prinicipal investigator, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304649
Record Dates: First submitted 2020-06-28; First posted 2020-07-14 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Optic Neuropathy
MeSH Terms: conditions — Optic Nerve Diseases | interventions — Erythropoietin

STUDY DESIGN:
Intervention Model Description: The study included 20 patients diagnosed as late onset optic neuropathy that are attending Alexandria main university hospital.
  All patients underwent initially assessment of visual acuity, color vision, pupil reaction ,funduscopy and electrophysiological tests ( pattern visual evoked potential and pattern electroretinogram in both eyes to use data of the normal fellow eye as patients' internal control). Systemic erythropoietin injections (eprax 10000 IU subcutaneous twice daily for three days). Follow up after one month and three months by recording visual acuity and electro physiological studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic erythropoietin injections (Experimental): 20 patients diagnosed as late onset optic neuropathy that were attending Alexandria main university hospital.Systemic erythropoietin injections (eprax 10000 IU subcutaneous twice daily for three days).
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: erythropoietin — Systemic erythropoietin injections (eprax 10000 IU subcutaneous twice daily for three days).

SUMMARY:
This study aimed to investigate the therapeutic effect of subcutaneous erythropoietin in the management of late stage optic neuropathy.

DETAILED DESCRIPTION:
Injury of the optic nerve or optic neuropathy is one of the most common causes of vision loss. This study aimed to investigate the therapeutic effect of subcutaneous erythropoietin in the management of late stage optic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with late stage optic neuropathy (1 month to 12 months after onset of optic neuropathy due to late referral of the cases)

Exclusion Criteria:

* Patients with perforating ocular injuries were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Assessment of visual acuity | 3 months
  Visual acuity using appropriate charts for assessment then convert into log of the minimum angle of resolution (logMAR) units to provide a numeric scale of visual acuity
Flash visual-evoked potentials | 3 months
  Flash VEP to detect amplitude reduction and latency in the optic nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Mai ElBahwash, PhD, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No